CLINICAL TRIAL: NCT02666846
Title: A Randomised, Double Blind, Cross Over Clinical Study in Healthy Human Volunteers to Assess the Efficacy and Safety of Three Different Topical Analgesics (DCF100, TIB200 And SPR300) Versus in a Model of UV-Induced Inflammatory Pain
Brief Title: Assess the Efficacy and Safety in Volunteers of DCF100, TIB200 and SPR300 vs. Placebo and Control(s) in a UV Pain Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Futura Medical Developments Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM52
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: UVB Pain Model; PK; Topical; NSAIDs
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Diclofenac; methyl salicylate; Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Cohort 1: TIB200 gel 10% (Experimental): All Cohort 1 participants: TIB200 gel (10%, w/w ibuprofen)
  Interventions: Drug: Ibuprofen
- Cohort 1: Nurofen gel 10% (Active Comparator): All Cohort 1 participants: Nurofen Max Strength gel (10%, w/w ibuprofen)
  Interventions: Drug: Ibuprofen
- Cohort 1: Nurofen tablets (Active Comparator): All Cohort 1 participants: Nurofen oral tablets (2 x 400 mg ibuprofen)
  Interventions: Drug: Ibuprofen
- Cohort 1: TIB200 Placebo gel (Placebo Comparator): All Cohort 1 Participants: TIB200 matching placebo gel
  Interventions: Drug: Placebo
- Cohort 2: DCF100 gel 2% (Active Comparator): All Cohort 2 Participants: DCF100 gel (2% w/w diclofenac)
  Interventions: Drug: Diclofenac
- Cohort 2: DCF100 gel 4% (Experimental): All Cohort 2 Participants: DCF100 gel (4% w/w diclofenac)
  Interventions: Drug: Diclofenac
- Cohort 2: Voltaren gel 2% (Active Comparator): All Cohort 2 Participants: Voltaren Emulgel (2% diclofenac)
  Interventions: Drug: Diclofenac
- Cohort 2: Voltarol oral tablet (Active Comparator): All Cohort 2 Participants: Voltarol oral tablet (50 mg - diclofenac)
  Interventions: Drug: Diclofenac
- Cohort 2: DCF100 Placebo gel (Placebo Comparator): All Cohort 2 Participants: DCF100 matching placebo gel
  Interventions: Drug: Placebo
- Cohort 3: SPR300 gel (15%:7%) (Active Comparator): All Cohort 3 Participants: Methyl-salicylate / Menthol, SPR300 gel (15%:7%, w/w; ratio of Methylsalicylate / Menthol)
  Interventions: Drug: Methyl-salicylate / Menthol
- Cohort 3: SPR300 Placebo gel (Placebo Comparator): All Cohort 3 Participants: SPR300 matching placebo gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen
  Other Names: TIB200 gel 10%, Nurofen gel 10%, Nurofen tablets
  Arms: Cohort 1: Nurofen gel 10%; Cohort 1: Nurofen tablets; Cohort 1: TIB200 gel 10%
Drug: Diclofenac
  Other Names: DCF100 gel 2%, DCF100 gel 4%, Voltaren gel 2%, Voltaren oral tablet
  Arms: Cohort 2: DCF100 gel 2%; Cohort 2: DCF100 gel 4%; Cohort 2: Voltaren gel 2%; Cohort 2: Voltarol oral tablet
Drug: Methyl-salicylate / Menthol
  Other Names: SPR300 gel (15%/7%)
  Arms: Cohort 3: SPR300 gel (15%:7%)
Drug: Placebo
  Other Names: TIB200 placebo gel, DCF100 placebo gel and SPR300 placebo gel
  Arms: Cohort 1: TIB200 Placebo gel; Cohort 2: DCF100 Placebo gel; Cohort 3: SPR300 Placebo gel

SUMMARY:
This is a randomised, double blind, cross over clinical study in healthy human volunteers (including pharmacokinetic [PK] sampling and laser Doppler assessment of local blood flow in a subset of up to 6 subjects per cohort of 20) to assess the efficacy and safety of three different topical analgesics (DCF100, TIB200 and SPR300) versus placebo and active control(s) in a model of UV-induced inflammatory pain.

DETAILED DESCRIPTION:
This is a randomised, double blind, cross over clinical study in healthy human volunteers, including pharmacokinetic (PK) sampling and laser Doppler assessment of local blood flow in a subset of up to 6 subjects per cohort, to assess the efficacy and safety of three different topical analgesics (DCF100, TIB200 and SPR300) versus placebo and active control(s) in a model of UV-induced inflammatory pain. The study will consist of 3 cohorts of subjects (n=20 subjects per cohort). Subjects of each cohort will receive test and reference products (no reference product for Cohort 3) of one investigational medicinal product (IMP) and a placebo.

Test Products:

Cohort 1: Ibuprofen, TIB200 gel (10%, w/w) Cohort 2: Diclofenac, DCF100 gel (2% or 4%, w/w) Cohort 3: Methyl-salicylate and Menthol, SPR300 gel (15%:7%, w/w; ratio of Methylsalicylate to Menthol)

Reference Products:

Cohort 1: Ibuprofen, Nurofen Max Strength gel (10%, w/w), Ibuprofen, Nurofen, oral tablet (400 mg) Cohort 2: Voltaren Emulgel (2%), Voltarol oral tablet (50 mg)

Placebo:

All Cohorts:Test product matching vehicle gel.

Pharmacodynamic tests and PK blood draws will be performed at: pre-dose, 1, 2, 4, and 6 hours post dose for all treatment cohorts and treatment days (PK blood sampling in up to 6 subjects per cohort only).

Safety will be evaluated by the incidence of local and systemic treatment-emergent adverse events (TEAEs) reported after each treatment. Safety assessments will also include vital signs, 12-Lead Electrocardiograms (ECGs), laboratory tests and a physical examination at Screening and the Follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Were able to provide written informed consent.
2. Male between 18 and 65 years old, inclusive, at the time of screening.
3. Good general health as ascertained by detailed medical history and physical examination.
4. Body mass index (BMI) ≥18 and ≤29 kg/m2 (BMI = weight/height2), at the time of screening.
5. No clinically relevant abnormalities in 12-lead ECG as per PI's judgement, e.g., absence of cardiac rhythm disorder, in particular bradycardia (<40 beats per minute), conduction abnormalities such as atrioventricular block, absence of active ischemia (such as unstable angina pectoris) or recent myocardial infarction, no QTcF interval >450 milliseconds, no QRS complex ≥120 milliseconds, at Screening.
6. No clinically relevant abnormalities in results of laboratory tests as per PI's judgement; in particular, no significant liver impairment defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT) 1.5x upper limit of normal (ULN); no significant kidney impairment defined as serum creatinine 2x ULN; abnormal thyroid function as defined by thyroid-stimulating hormone (TSH) and total thyroxin (T4) (TSH within range 0.27 to 4.2 mIU/L, total T4 within range 59 to 154 nmol/L).
7. Had a skin type II or III (Fitz Patrick classification).
8. Non-smokers or ex-smokers for at least 6 months prior to the Screening Visit, as confirmed by a urine cotinine test.
9. Subjects were able to communicate well with the PI/designee. -

Exclusion Criteria:

1. History of hypersensitivity to the IMP or any of the excipients or to medicinal products with similar chemical structures.
2. Presence of any clinically relevant acute or chronic disease which could interfere with the subject safety during the study, expose the subject to undue risk, limit the biological sampling (e.g., blood collection), interfere with the absorption of the IMP (e.g., active dermatological conditions at the application sites, or ulcers, irritable bowel syndrome) or interfere with the study objectives.
3. Skin type I, IV, V or VI (Fitzpatrick Classification).
4. History of chronic pain symptoms (>6 months) or ongoing pain.
5. Any condition that required regular concomitant medication including herbal products, or predicted need of any concomitant medication from Screening Visit until the end of the study.
6. Intake of any medication including over the counter (OTC) medication (in particular any pain killers), herbal and dietary supplements such as St John's Wort, vitamins and minerals that could affect the outcome of the study, within 48 hours before the first administration of the investigational product and for the duration of the study.
7. Use of photosensitising medication, such as phenothiazines, tetracyclines, quinolones, sulphonamides, nalidixic acid, non-steroidal anti-inflammatories, furosemides, hydrochlorothiazides, fibrate, phytotherapeutic drugs (herbal supplements), phenothiazines, quinidines, psoralens and amiodarone within 4 weeks before the first UVB irradiation and for the duration of the study.
8. Any skin disease, acute or chronic (e.g., psoriasis vulgaris, neurodermatitis) or auto immune diseases associated with increased light sensitisation.
9. Any active dermatological conditions, local pigmentary disorders, body art (e.g., tattoos), or excessive hair growth at the lower back that might interfere with the study assessments or absorption of the IMP.
10. History of skin cancer (i.e., melanoma, squamous cell carcinoma or basal cell carcinoma).
11. History of conditions that increase risk for melanoma (e.g., dysplastic nevus [>5 nevi], xeroderma pigmentosum, Fanconi anaemia, Bloom's syndrome, Werner syndrome, Cockayne syndrome, trichothiodystrophy, or familial mole melanoma syndrome).
12. History of bleeding disorders, peptic ulceration or gastro intestinal bleeding, heart burn, cardiovascular disease, myocardial infarction or stroke.
13. Inability to give reproducible HPPT ratings on naïve skin at screening, (defined as HPTT test re-test difference ≥1.0 °C)
14. Heat pain perception threshold <40°C or >51°C on naïve skin at Screening.
15. Supine systolic blood pressure (SBP) <90 mmHg or >140 mmHg, or supine diastolic blood pressure (DBP) <50 mmHg or >90 mmHg after 5 minutes supine, at the Screening Visit.
16. Positive test results for HBsAg, HCVAb or HIV-1 and/or -2 antibodies at Screening.
17. Excessive use of caffeine-containing beverages exceeding 500 mg caffeine/day (5 cups of coffee) and the inability to refrain from the use of caffeine-containing beverages during confinement in the Clinical Unit.
18. Excessive alcohol consumption (regular alcohol intake ≥21 units per week). Use of alcohol 48 hours before any study visit, as confirmed by urine alcohol testing at Screening, Day -2, and with any additional tests at the discretion of the PI.
19. History in the last year or presence of drug addiction (positive urine drug screen) at Screening and Day -2.
20. Presence or history of alcohol abuse in the last year, as confirmed by subject's general practitioner (GP).
21. Blood donation within 8 weeks before the first IMP administration.
22. Participation in another study with an experimental drug within 3 months before the first dosing day.
23. Any psychological, emotional problems, any disorder or resultant therapy that was likely to invalidate informed consent, or limited the ability of the subject to comply with the protocol requirements.
24. Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for Follow-up visits and improbability of completing the clinical study.
25. Planned surgery, dental procedure, or hospitalisation from the Screening Visit until the end of the study.
26. Inability to give written informed consent or to comply fully with the protocol.
27. Subjects who, in the opinion of the PI, were considered unsuitable for any other reason.

    -

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBChB, Principal Investigator — PAREXEL Ltd.
Locations (1):
- PAREXEL EPCU Northwick Park, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Dosed on Days 1, 2 and 3): All Cohort 1 participants: Ibuprofen (day 1), TIB200 gel (10%, w/w) (Day 2) and TIB200 (placebo gel) (Day 3)
  (Follow up 7-9 days post last UVB irradiation)
  Ibuprofen: Single topical dose per 1.76 cm2 test site of: 22 microliters (μL) (20 ± l mg)* of TIB200 Gel (ibuprofen 10% w/w) (Test Gel) or 22 μL (20 ± l mg)* of matching placebo TIB200 Gel (placebo gel) or 22 μL (20 ± l mg)* of Nurofen Maximum Strength Gel (ibuprofen 10% w/w) (reference gel).
- Cohort 2 (Dosed on Days 1,2,3 and 4): All Cohort 2 Participants: Diclofenac, DCF100 gel (2% w/w) (day 1), DCF100 gel (4% w/w) (day 2), DCF100 gel (marching placebo) Day 3 and Voltarol® 12 Hour Emulgel® P 2.32% Gel (day 4)
  (Follow up 7-9 days post last UVB irradiation)
  Diclofenac: Subjects were randomised to receive 22 uL (20 ± l mg) DCF100 Gel (diclofenac 2% w/w) / DCF100 Gel (diclofenac 4% w/w) / Matching Placebo DCF100 Gel / Voltarol® 12 Hour Emulgel® P 2.32% Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 3 (Dosed on Days 1 and 2): All Cohort 3 Participants: Methyl-salicylate / Menthol, SPR300 gel (15%:7%, w/w; ratio of Methylsalicylate / Menthol) (day 1) and SPR300 (Matching Placebo) (day 2)
  Follow up visit between days 7-9 post last UVB irradiation
  Methyl-salicylate / Menthol: Subjects were randomised to receive 22 uL (20 ± l mg) SPR300 Gel / Matching Placebo SPR300 Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
Period: Overall Study
Arm/Group | Cohort 1 (Dosed on Days 1, 2 and 3) | Cohort 2 (Dosed on Days 1,2,3 and 4) | Cohort 3 (Dosed on Days 1 and 2)
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Cohort 1:
  Ibuprofen: Single topical dose per 1.76 cm2 test site of: 22 microliters (μL) (20 ± l mg)* of TIB200 Gel (ibuprofen 10% w/w) (Test Gel) or 22 μL (20 ± l mg)* of matching placebo TIB200 Gel (placebo gel) or 22 μL (20 ± l mg)* of Nurofen Maximum Strength Gel (ibuprofen 10% w/w) (reference gel) or Ibuprofen, Nurofen oral tablets (2 x 400 mg)
- Cohort 2:: Cohort 2:
  Diclofenac: Subjects were randomised to receive 22 uL (20 ± l mg) DCF100 Gel (diclofenac 2% w/w) / DCF100 Gel (diclofenac 4% w/w) / Matching Placebo DCF100 Gel / Voltarol® 12 Hour Emulgel® P 2.32% Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 3: Cohort 3:
  Methyl-salicylate / Menthol: Subjects were randomised to receive 22 uL (20 ± l mg) SPR300 Gel / Matching Placebo SPR300 Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2: | Cohort 3 | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 20 | 20 | 60
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 20 | 20

OUTCOME MEASURES:

1. Primary Outcome: Heat Pain Tolerance Test (HPTT) Measured the Point at Which the Heat Became Painful - Degrees Centigrade -
Description: To assess the pharmacodynamic effect by Heat Pain Tolerance Test (HPTT) which measured the point at which the heat became painful (degrees centigrade) of three topical analgesics, DCF100, TIB200, and SPR300 versus topical placebo and active topical reference products in a model of UV-induced inflammatory pain.
Time Frame: 15 minutes before to 6 hours post administration
Measure: Mean (Standard Deviation); unit: Degrees Centigrade
Groups:
- Cohort 1: TIB200 Gel 10%: Cohort 1: Ibuprofen, TIB200 gel (10%, w/w)
  Ibuprofen: Single topical dose per 1.76 cm2 test site of: 22 microliters (μL) (20 ± l mg)* of TIB200 Gel (ibuprofen 10% w/w) (Test Gel) or 22 μL (20 ± l mg)* of matching placebo TIB200 Gel (placebo gel) or 22 μL (20 ± l mg)* of Nurofen Maximum Strength Gel (ibuprofen 10% w/w) (reference gel).
- Cohort 1: Nurofen Gel 10%: Cohort 1: Ibuprofen, Nurofen Max Strength gel (10%, w/w)
  Ibuprofen: Single topical dose per 1.76 cm2 test site of: 22 microliters (μL) (20 ± l mg)* of TIB200 Gel (ibuprofen 10% w/w) (Test Gel) or 22 μL (20 ± l mg)* of matching placebo TIB200 Gel (placebo gel) or 22 μL (20 ± l mg)* of Nurofen Maximum Strength Gel (ibuprofen 10% w/w) (reference gel).
- Cohort 1: Nurofen Tablets: Cohort 1: Ibuprofen, Nurofen oral tablets (2 x 400 mg)
  Ibuprofen: Single topical dose per 1.76 cm2 test site of: 22 microliters (μL) (20 ± l mg)* of TIB200 Gel (ibuprofen 10% w/w) (Test Gel) or 22 μL (20 ± l mg)* of matching placebo TIB200 Gel (placebo gel) or 22 μL (20 ± l mg)* of Nurofen Maximum Strength Gel (ibuprofen 10% w/w) (reference gel).
- Cohort 1: TIB200 Placebo Gel: Cohort 1: TIB200 matching placebo gel
  Placebo: The placebo gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 2: DCF100 Gel 2%: Cohort 2: Diclofenac, DCF100 gel (2% w/w)
  Diclofenac: Subjects were randomised to receive 22 uL (20 ± l mg) DCF100 Gel (diclofenac 2% w/w) / DCF100 Gel (diclofenac 4% w/w) / Matching Placebo DCF100 Gel / Voltarol® 12 Hour Emulgel® P 2.32% Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 2: DCF100 Gel 4%: Cohort 2: Diclofenac, DCF100 gel (4% w/w)
  Diclofenac: Subjects were randomised to receive 22 uL (20 ± l mg) DCF100 Gel (diclofenac 2% w/w) / DCF100 Gel (diclofenac 4% w/w) / Matching Placebo DCF100 Gel / Voltarol® 12 Hour Emulgel® P 2.32% Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 2: Voltaren Gel 2%: Cohort 2: Diclofenac, Voltaren Emulgel (2%)
  Diclofenac: Subjects were randomised to receive 22 uL (20 ± l mg) DCF100 Gel (diclofenac 2% w/w) / DCF100 Gel (diclofenac 4% w/w) / Matching Placebo DCF100 Gel / Voltarol® 12 Hour Emulgel® P 2.32% Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 2: Voltarol Oral Tablet: Cohort 2: Diclofenac, Voltarol oral tablet (50 mg)
  Diclofenac: Subjects were randomised to receive 22 uL (20 ± l mg) DCF100 Gel (diclofenac 2% w/w) / DCF100 Gel (diclofenac 4% w/w) / Matching Placebo DCF100 Gel / Voltarol® 12 Hour Emulgel® P 2.32% Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 2: DCF100 Placebo Gel: Cohort 2: DCF100 matching placebo gel
  Placebo: The placebo gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 3: SPR300 Gel (15%:7%): Cohort 3: Methyl-salicylate / Menthol, SPR300 gel (15%:7%, w/w; ratio of Methylsalicylate / Menthol)
  Methyl-salicylate / Menthol: Subjects were randomised to receive 22 uL (20 ± l mg) SPR300 Gel / Matching Placebo SPR300 Gel. The gels were administered topically on two test sites on the lower back of the subject, each 1.76cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
- Cohort 3: SPR300 Placebo Gel: Cohort 3: SPR300 matching placebo gel
  Placebo: The placebo gels were administered topically on two test sites on the lower back of the subject, each 1.76 cm2 in size. The two test sites were UVB irradiated on the previous day, between 22 and 26 hours (24 ± 2 hours) before dosing.
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 1: TIB200 Placebo Gel | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 2: DCF100 Placebo Gel | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Degrees Centigrade | 0.3635 (1.0277) | 0.7358 (1.0277) | 0.0887 (0.9024) | -0.1983 (0.4616) | 0.6679 (1.0657) | 0.8722 (1.0430) | 0.7978 (0.9780) | 0.6835 (0.7344) | 0.1688 (0.7231) | 0.3934 (1.2384) | -0.0123 (1.0103)

2. Primary Outcome: Intensity of the UVB-induced Erythema (Determined by Assessment of Skin Blood Flow by Laser Doppler Imaging [Flux Units])
Description: Intensity of the Ultra Violet B radiation (UVB)-induced erythema (determined by assessment of skin blood flow by laser Doppler imaging [flux units], up to 8 subjects per cohort) - Change from baseline
Time Frame: 15 minutes before to 6 hours post administration
Measure: Least Squares Mean (Standard Deviation); unit: Laser doppler imaging (Flux Units)
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 1: TIB200 Placebo Gel | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 2: DCF100 Placebo Gel | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Laser doppler imaging (Flux Units) | -313.3879 (105.7042) | -171.5589 (96.6485) | -262.0693 (88.5449) | -95.3974 (81.4103) | -228.3016 (183.2260) | -278.1918 (103.7333) | -198.1408 (133.2886) | -198.1408 (211.2754) | -45.376 (104.4476) | 12.2265 (111.1065) | 67.3931 (91.092)

3. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax), time corresponding to occurrence of Cmax (tmax) (up to 6 subjects per cohort only) laser Doppler imaging [flux units], up to 6 subjects per cohort)
Time Frame: 15 minutes before and 1, 2, 4 and 6 hours post administration
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/ml | 11.5 (14) | 5.15 (8.1) | 29900 (5490) | 0 (0) | 0 (0) | 0 (0) | 772 (468) | 0 (0) | 0 (0)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve
Description: Area under the concentration vs. time curve from time zero to 6 hours (AUC0-6h) (up to 6 subjects per cohort only) laser Doppler imaging [flux units], up to 6 subjects per cohort)
Time Frame: 15 minutes before and 1, 2, 4 and 6 hours post administration
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
h*ng/ml | 47.7 (64.3) | 19.9 (33.7) | 90000 (15400) | 0 (0) | 0 (0) | 0 (0) | 1030 (463) | 0 (0) | 0 (0)

5. Secondary Outcome: Number of Recorded Abnormal Clinical Assessments
Description: Laboratory assessments - standard clinical trial assessments for clinical chemistry and haematology
  Listing of individual laboratory measurements by subjects and evaluation of each laboratory parameter
Time Frame: Estimated study duration for each subject will be approximately 6 weeks
Measure: Number; unit: Assessments
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 1: TIB200 Placebo Gel | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 2: DCF100 Placebo Gel | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Assessments | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Physical Exams to Ensure Safety and Well Being of the Subjects
Description: Physical examinations - including assessments of the application site. examination.
Time Frame: Estimated study duration for each subject will be approximately 6 weeks
Measure: Number; unit: Abnormalities
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 1: TIB200 Placebo Gel | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 2: DCF100 Placebo Gel | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Abnormalities | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Adverse Events (AEs)
Description: Local and systemic Adverse Events (AEs).
Time Frame: Estimated study duration for each subject will be approximately 6 weeks
Measure: Number; unit: Events
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 1: TIB200 Placebo Gel | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 2: DCF100 Placebo Gel | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Events | 5 | 5 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 3 | 1

8. Secondary Outcome: To Determine Vital Signs and Electrocardiograms (ECGs) That Were Abnormal to Ensure Safety and Well Being of the Subjects
Description: To determine Vital Signs and Electrocardiograms (ECGs) that were abnormal to ensure safety and well being of the subjects
Time Frame: Estimated study duration for each subject will be approximately 6 weeks
Measure: Number; unit: Abnormal readings
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 1: TIB200 Placebo Gel | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 2: DCF100 Placebo Gel | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Abnormal readings | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: All AE's were reported as this was a phase 1 study
  The threshold for reporting was therefore greater than 0%
Arm/Group | Cohort 1: TIB200 Gel 10% | Cohort 1: Nurofen Gel 10% | Cohort 1: Nurofen Tablets | Cohort 1: TIB200 Placebo Gel | Cohort 2: DCF100 Gel 2% | Cohort 2: DCF100 Gel 4% | Cohort 2: Voltaren Gel 2% | Cohort 2: Voltarol Oral Tablet | Cohort 2: DCF100 Placebo Gel | Cohort 3: SPR300 Gel (15%:7%) | Cohort 3: SPR300 Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 5/20 | 1/20 | 1/20 | 1/20 | 1/20 | 0/20 | 2/20 | 0/20 | 3/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: TIB200 Gel 10% (N=20) | Cohort 1: Nurofen Gel 10% (N=20) | Cohort 1: Nurofen Tablets (N=20) | Cohort 1: TIB200 Placebo Gel (N=20) | Cohort 2: DCF100 Gel 2% (N=20) | Cohort 2: DCF100 Gel 4% (N=20) | Cohort 2: Voltaren Gel 2% (N=20) | Cohort 2: Voltarol Oral Tablet (N=20) | Cohort 2: DCF100 Placebo Gel (N=20) | Cohort 3: SPR300 Gel (15%:7%) (N=20) | Cohort 3: SPR300 Placebo Gel (N=20)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain Burning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequency of Micturation Increased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft Stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Commom Cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythematous Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No